## INFORMED CONSENT FORM

**Tittle**: Inhibitory Control Training for the Treatment of Excess Weight: Behavioral, Cognitive and Anthropometric Changes (InhibeT)

Code:

Date: September 2024

## INFORMATION SHEET

STUDY NAME: Inhibitory Control Training for the Treatment of Excess Weight: Behavioral, Cognitive and Anthropometric Changes (InhibeT)

Responsible researchers: Raquel Vilar López and Alfonso Caracuel Romero Mind, Brain and Behavior Research Center of the University of Granada Email:

rvilar@ugr.es; acaracuel@ugr.es

Please read this information carefully: Your voluntary participation in a research project is requested. Before participating in the study, please read the information we provide below and ask as many questions as you need to ensure that you understand what your participation entails.

# Information about the study and your participation in itWhat are the objectives of the study?

The objective of this study is to determine the effectiveness of a program for the treatment of excess weight. The present study uses the Food Trainer App to investigate whether it improves the results of cognitive training aimed at the adherence of healthy habits and weight loss.

Additionally, we aim to better understand the relationship between measures related to weight, and their association with other cognitive measures will be determined (food evaluation, frequency of physical exercise, decision making, inhibition, working memory, flexibility)

#### Where is the study carried out?

This study is directed by Raquel Vilar López and Alfonso Caracuel Romero, and their collaborating team. The study will be online from the Mind, Brain and Behavior Research Center (CIMCYC), belonging to the University of Granada, and located on the La Cartuja Campus (between the faculties of Psychology and Pharmacy).

#### What procedures will I carry out?

This study has an evaluation part and an intervention part.

In the evaluation you will carry out different tasks (pencil and paper and/or through the computer and mobile phone) with which we can learn different aspects related to your way of eating and psychological aspects (such as impulsivity and personality), in addition to your weight and height, in a session of about 120 minutes.

These evaluations will be carried out at three time points: before starting the intervention sessions, the week after finishing said sessions, and in the follow-up that we will carry out 3 months after finishing the intervention.

In the interventions itself you will carry out inhibitory control training with your mobile phone for 10 minutes.

# Are there any drawbacks to participating in the study?

The different evaluation sessions and cognitive tasks do not present any inconvenience for the participants, beyond the mental fatigue that some people may feel from carryingout these types of activities.

#### Is there any benefit from participating in the study?

Participation in the study could provide you with benefits related to the improvement of certain aspects of impulsivity, and therefore could help you reduce excess weight.

There is no financial compensation. You have the right to receive a report of your evaluation performance.

In addition, your participation will provide scientific knowledge that will contribute to improving the design of treatments for excess weight.

### Confidentiality

The personal data required (name, age, sex, health data and habits collected in the evaluation) are those necessary to cover the objectives of the study. All data obtained will be used solely and exclusively for the objectives of the studyand will be treated by the research team in a completely confidential manner. The results derived from this study can be published in a scientific journal or conference, always maintaining anonymity and confidentiality. Any personally identifiable information will be kept and processed securely. Data may only be shared in repositories for scientific purposes in a format that guarantees the maintenance of anonymity.

During the completion of the study, you may at any time exercise your right of access, rectification, cancellation and opposition to your data before the responsible researcher, as established by royal decree 1720/2007, Organic Law 3/2018 on the Protection of Personal Data and guarantee of digital rights, and the European directive 2002/58/EC. You can obtain additional information on your rights regarding the processing of your data at <a href="http://secretariageneral.ugr.es/pages/proteccion\_datos/derechos">http://secretariageneral.ugr.es/pages/proteccion\_datos/derechos</a>, and by contacting the email address: protecciondedatos@ugr.es

#### **Study Participation Agreement**

This sheet contains information so you can decide if you want to participate in this study. If you have any questions that remain unanswered, please ask the study manager before signing this form. You can contact the main researchers of the project, Raquel Vilar López and Alfonso Caracuel Romero, through email <a href="mailto:rvilar@ugr.es">rvilar@ugr.es</a> and <a href="mailto:acaracuel@ugr.es">acaracuel@ugr.es</a> or by phone 958241982 and 958242948.

Participation in this study is voluntary, and you will have the possibility to revoke your consent at any time and without having to give explanations. You do not have to participate in the study if you do not want to. If you ultimately decide to participate, you will receive a copy to keep this information and another to sign giving your consent.

#### INFORMED CONSENT SHEET

**Project title:** Inhibitory Control Training for the Treatment of Excess Weight: Behavioral, Cognitive and Anthropometric Changes (InhibeT)

PROFESSIONALS INVOLVED IN THE INFORMATION AND/OR CONSENT PROCESS:

The following professionals declare that the information regarding participation in the project has been explained:

Raquel Vilar López and Alfonso Caracuel Romero

Mind, Brain and Behavior Research Center of the University of GranadaID: 46898000B and 52363377J

#### 1. CONSENT TO PARTICIPATE IN THE STUDY:

| I, Mr./Mrs. (name and surname) | |
|--------------------------------|---------|
| with <b>ID number</b> | <u></u> |

I declare under my responsibility that I have read and understood the Information sheet, a copy of which has been given to me.

I have received sufficient information about my participation in the project, about the use of my persnal data and associated information.

I have been able to ask questions about the information received and speak with the indicated professional, who has resolved all the doubts I have raised.

I understand that my participation is voluntary.

I understand that all my data will be treated confidentially, according to Regulation (EU) 2016/679 General Data Protection and Organic Law 3/2018 on the Protection of Personal Data and Guarantee of Digital Rights.

I understand that I can withdraw from the study:

- Whenever you want.
- Without having to give explanations.
- Without this affecting me in any way.

| J | i give my c | consent to | or the cli | nical data | a to be | treated | in the | tollowing | manner: |
|---|---|---|---|---|---|---|---|---|---|

| $\Box$ Encrypted (they will be identified with a code that protects my identity, making it possible to link them back to me) |
|---|
| I authorize you to contact me later: |
| □ YES |
| □ NO |
| If so, please indicate the means to do so: |
| ☐ Telephone: (insert number) |
| ☐ Email: (insert address) |
| Others: (identify) |

| I wish to establish restr | ictions regarding the use of th | e sample, so that it is not used |
|---|---|---|
| in: | | |
| I authorize receiving into of my family members | C | nd data relevant to my health andthat |
| Check what applies: | | |
| □ YES | | |
| □ NO | | |
| I know that I can revok | e, at any time, the consent gra | nted in this document. |
| OnSIGNATURE | , onof | , 20 |